CLINICAL TRIAL: NCT04825769
Title: A Randomized Controlled Trial of Low-dose Single-wavelength Red Light in the Decrease of Myopia Incidence Rate in the Setting of School.
Brief Title: Red Light Intervention for Myopia Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SHYB2021001
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Myopia
Keywords: Children and adolescents; Myopia; Prevention and control; Red light
MeSH Terms: conditions — Myopia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Red light irradiation was conducted at school from Monday to Friday and at home everyday in summer and winter holiday twice a day for 3 minutes per time, with an interval of 4 hours
  Interventions: Device: LLLT（Low Level Laser Therapy）
- Control (No Intervention): No intervention

INTERVENTIONS:
Device: LLLT（Low Level Laser Therapy） — 2 times a day, 3 minutes each time, with an interval of more than 4 hours. During the semester: From Monday to Friday, set up an intervention room in the school; For winter and summer vacation: everyday at home
  Arms: Intervention

SUMMARY:
To explore the effectiveness of using low-intensity single-wavelength red light to prevent myopia in schoolchildren, and to provide a feasible scheme for reducing the incidence of myopia.

ELIGIBILITY:
Inclusion Criteria:

* Students of grade 1-4 in the participating schools;
* Students' eyes have no myopia, that is the cycloplegic spherical equivalent（SE） >-0.50D, and at least one eye accords with the pre-myopic state, that is -0.50D <cycloplegic SE≤0.50D;
* Students whose mother and/or father are in myopia status (SE < -3.0D for either of eyes);
* Students whose parents sign informed consent and agree to let their kids participate in baseline screen and follow-up examinations and surveys.

Exclusion Criteria:

* Students whose parents do not sign informed consent;
* Students who have strabismus and/or other binocular vision abnormality;
* Students who have other eye diseases and/or systematic diseases;
* Students who have DC <=-1.5D;
* Students whose difference of SE between the two eyes >=1.5D;
* Students who meet the standards with which investigators and study physicians think it is not appropriate to enroll.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
One-year cumulative incidence of myopia (%) in the intervention group and the control group. | 1 year
  Myopia is defined as the cycloplegic spherical equivalent of either eye ≤-0.5D

SECONDARY OUTCOMES:
The progress of spherical equivalent(SE,D) of children in intervention group and control group. | 1 year
  The spherical equivalent(SE,D) will be measured by autorefractor(KR-8900, Topcon).
The progress of axial length of children in intervention group and control group. | 1 year
  The axial length will be measured using IOLMaster.
The progress of choroidal thickness in children in pre-myopia state in intervention group and control group. | 1 year
  The choroidal thickness will be measured using SS-OCT.
The change of uncorrected visual acuity (UCVA) of children in intervention group and control group. | 1 year
  The uncorrected visual acuity (UCVA) will be measured using a mounted and illuminated E chart of the Early Treatment Diabetic Retinopathy study (ETDRS) charts.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangui He, Study Director — Shanghai Eye Disease Prevention and Treatment Center
Locations (1):
- Xiangui He, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He X, Wang J, Zhu Z, Xiang K, Zhang X, Zhang B, Chen J, Yang J, Du L, Niu C, Leng M, Huang J, Liu K, Zou H, He M, Xu X. Effect of Repeated Low-level Red Light on Myopia Prevention Among Children in China With Premyopia: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e239612. doi: 10.1001/jamanetworkopen.2023.9612. PMID 37099298

DOCUMENTS (3):
  • Study Protocol (2021-03-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT04825769/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT04825769/SAP_001.pdf
  • Informed Consent Form (2021-03-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT04825769/ICF_002.pdf